CLINICAL TRIAL: NCT00307957
Title: Pillar Palatal Implant System Multi-Institutional, Randomized Placebo-Controlled Study for Obstructive Sleep Apnea
Brief Title: Study to Determine the Effectiveness of Pillar Palatal Implants to Treat Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Medtronic Xomed, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-08-14-1
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Daytime Sleepiness; Pillar Palatal Implants
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence

INTERVENTIONS:
Device: Pillar Palatal Implants

SUMMARY:
The Pillar palatal implant procedure is a minimally invasive and commercially available treatment for mild to moderate obstructive sleep apnea (OSA) in the United States and Europe. The implants are placed into the soft area in the roof of the mouth providing support to the soft palate. This research is being done to compare daytime sleepiness and sleep related quality of life after palatal implants.

DETAILED DESCRIPTION:
Patients will be enrolled into the study based on sleep study results, a physical exam and inclusion/exclusion criteria. Once enrolled, patients are randomized into either the Pillar palatal implant group or a placebo/sham group.

In both cases, patients come into the office for placement of the implants. This is an outpatient procedure. Patients are followed at one week, one month and 3 months. At each follow-up visit, patients will undergo a physical exam and complete questionnaires related to sleep and quality of life. Patients will also undergo reaction time testing on hand-held device similar to a pocket video game. At the three month visit, patients will return to the sleep lab for another sleep study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Body Mass Index equal to 32 or less
* Apnea-Hypopnea Index greater than/equal to 10 and less than/equal to 30
* Symptoms of daytime sleepiness

Exclusion Criteria:

* Septal deviation or nasal obstruction
* Nasal polyps
* Severe seasonal allergies
* Soft palate length insufficient to accommodate implants
* Fujita Modified Mallampati Class 3
* Large tonsils
* Lingual tonsil hypertrophy
* Hypopharyngeal obstruction
* Previous pharyngeal surgery
* Previous upper respiratory tract cancer or radiation therapy
* Active respiratory tract infection
* Dysphagia or speech disorder
* Neurologic disorder
* Unstable psychiatric disorder
* Pregnant or breastfeeding
* History of falling asleep driving or MVA due to sleepiness
* Currently on CPAP therapy or other device for OSA
* Other sleep disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Daytime Sleepiness (ESS)
Apnea/Hypopnea Index (AHI)

SECONDARY OUTCOMES:
Sleep Related Quality of Life (FOSQ)
Reaction Time Testing (PVT)
Other polysomnographic parameters (AI, HI, RERArl, Arl, LSat)

CONTACTS AND LOCATIONS:
Overall Officials: David L Steward, MD, Principal Investigator — University Ear, Nose and Throat Specialists
Locations (3):
- United States (3):
  - University of Indiana Medical Center, Indianapolis, Indiana
  - University Ear, Nose and Throat Specialists, Cincinnati, Ohio
  - Department of OTO-HNS Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Manufacturer's website for more information on Pillar Implants — http://www.restoremedical.com